CLINICAL TRIAL: NCT05675098
Title: Effect of Central Nervous System Stimulants on Physical Function in Children With Cerebral Palsy: A Pilot Randomized Controlled Trial
Brief Title: Central Nervous System Stimulants and Physical Function in Children With Cerebral Palsy
Acronym: CP
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Kuwait University (Other)
Responsible Party: Principal Investigator, Dr. Anwar Amutairi, Assistant Professor, Kuwait University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IRB-2157/2022
Record Dates: First submitted 2022-12-13; First posted 2023-01-09 (Actual); Last update posted 2023-03-08 (Actual); Status verified 2023-03

CONDITIONS: Neurodevelopmental Disorders; Cerebral Palsy
Keywords: methylphenidate; Modafinil; physical therapy; motor performance; spasticity; physical function
MeSH Terms: conditions — Neurodevelopmental Disorders; Cerebral Palsy; Muscle Spasticity | interventions — Methylphenidate; Modafinil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Methylphenidate (Experimental): Participants in this group will receive 2.5mg Methylphenidate and 100mg placebo (Modafinil shape) in addition to physical therapy program
  Interventions: Drug: Methylphenidate
- Modafinil (Experimental): Participants in this group will receive 100mg Modafinil and 2.5mg placebo (Methylphenidate shape) in addition to physical therapy program
  Interventions: Drug: Modafinil
- Placebo (Placebo Comparator): Participants in this group will receive 2.5mg placebo (Methylphenidate shape) and 100mg placebo (Modafinil shape) in addition to physical therapy program
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Methylphenidate — This medication is a psychostimulant medication and is usually prescribed for individuals with Attention-Deficit/Hyperactivity Disorder to manage ADHD behavioral symptoms
  Other Names: Ritalin
  Arms: Methylphenidate
Drug: Modafinil — This medication is a Central Nervous System stimulant and is usually used to treat neurological conditions, including Narcolepsy
  Other Names: Provigil
  Arms: Modafinil
Other: Placebo — Participant will receive placebo tablets (Methylphenidate and Modafinil shape)
  Other Names: Control
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine the effects of Central Nervous System Stimulants, represented by Methylphenidate and Modafinil, compared to placebo control on motor performance in children with Cerebral Palsy. This study will be a triple-masked study per the American Academy of Neurology guidelines for clinical trials.

DETAILED DESCRIPTION:
Cerebral Palsy (CP) is a neurological disorder that commonly cause disability and limit physical function in children, and this disability persists into adulthood. There are several treatment options for motor impairments associated with CP, including oral medications (diazepam or related benzodiazepines, baclofen, dantrolene, and tizanidine hydrochloride), intraspinal infusion (baclofen), paralyzing agents (Botulinum toxin), and surgical interventions (dorsal rhizotomy). However, these interventions have drawbacks that could impact their benefits, such as drowsiness with oral medications and permanent change in muscle tone with the rhizotomy surgery. Other rehabilitation interventions showed significant improvements in motor function such as constraint-induced movement therapy (CIMT) and strength training. A few researchers attempted using central nervous system stimulants (i.e., Modafinil [Provigil]) off-label for improving motor control and reducing spasticity in children with CP. Another medication that has been used for motor impairments is Methylphenidate (MPH), also a central nervous system stimulant. However, this medication was used for improving muscle tone and motor performance in children with Attention-deficit/Hyperactivity Disorder (ADHD), but not in children with CP. MPH is useful for children with combined CP and ADHD and showed beneficial results for ADHD symptoms and behavioral outcomes with minimal side effects. Therefore, the purpose of this pilot randomized controlled trial (RCT) is to examine the effects of Central Nervous System (CNS) stimulants (Modafinil and MPH) vs. placebo in addition to physical therapy intervention on gross motor function and spasticity in children with CP.

ELIGIBILITY:
Inclusion Criteria:

* Children diagnosed with spastic diplegic or quadriplegic CP by a physician.
* Children aged between 7-12 years old.
* Children with CP classified as level I & II based on the gross motor function classification system (GMFCS).
* Children with CP that are receiving physical therapy for ≥ 3 months.

Exclusion Criteria:

* Children that had a seizure attack in the past 6 months
* Children that have been diagnosed with attention deficit/ hyperactivity disorder (ADHD)
* Children that had any surgery within the last 6 months
* Children that has lower-extremity contractures determined by the passive range of motion (hips, knees, and ankles)
* Children that use medications that interfere with spasticity (e.g., Baclofen)

Ages: 7 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2023-05-01 (Estimated); Primary Completion 2025-02-01 (Estimated); Study Completion 2027-02-01 (Estimated)

PRIMARY OUTCOMES:
Gross motor function measure (GMFM) | Baseline, 6 weeks, 12 weeks, and 24 weeks after intervention
  To determine changes in functional motor abilities.
Modified Ashworth Scale (MAS) | Baseline, 6 weeks, 12 weeks, and 24 weeks after intervention
  To determine changes in spasticity

SECONDARY OUTCOMES:
Body height | Baseline, 6 weeks, 12 weeks, and 24 weeks after intervention
  To determine body height
Timed up and go (TUG) | Baseline, 6 weeks, 12 weeks, and 24 weeks after intervention
  To assess dynamic balance
Five times sit to stand test (5x Sit-To-Stand Test /5XSST) | Baseline, 6 weeks, 12 weeks, and 24 weeks after intervention
  To assess the change in functional strength
Modified clinical test for sensory interaction of balance (MCTSIB) | Baseline, 6 weeks, 12 weeks, and 24 weeks after intervention
  To assess static balance
Ten-meter walk test (10MWT) (normal pace) | Baseline, 6 weeks, 12 weeks, and 24 weeks after intervention
  To assess change in gait speed
2-Minutes Walking Test (normal pace) | Baseline, 6 weeks, 12 weeks, and 24 weeks after intervention
  To determine changes in fatigue
The University of California, San Diego Shortness of Breath Questionnaire (UCSDSOBQ) | Baseline, 6 weeks, 12 weeks, and 24 weeks after intervention
  To determine changes in respiratory function
Body weight | Baseline, 6 weeks, 12 weeks, and 24 weeks after intervention
  To determine body weight

CONTACTS AND LOCATIONS:
Overall Officials: Anwar B Almutairi, PT, PhD, Principal Investigator — Kuwait University
Locations (1):
- Physical Medicine and Rehabilitation Hospital, Kuwait City, Kuwait

IPD SHARING:
Plan to Share IPD: No
To be determined

REFERENCES:
- [Derived] Alotaibi M, Almutairi AB, Alhirsan S, Alkazemi A, Alharbi M, Alrashdi N, Taqi A, Alamiri B, Vogtle L, Alqahtani MM. Psychostimulant Medications for Physical Function and Spasticity in Children With Cerebral Palsy: Protocol for a Randomized Controlled Trial. JMIR Res Protoc. 2024 Mar 5;13:e53728. doi: 10.2196/53728. PMID 38441919